CLINICAL TRIAL: NCT01261728
Title: Phase II Study of Gemcitabine and Cisplatin as Neoadjuvant Chemotherapy in Patients With High-Grade Upper Tract Urothelial Carcinoma
Brief Title: Gemcitabine and Cisplatin as Neoadjuvant Chemotherapy in Patients With High-Grade Upper Tract Urothelial Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Mayo Clinic (Other); Hartford Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-208
Record Dates: First submitted 2010-12-15; First posted 2010-12-16 (Estimated); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Urothelial Carcinoma
Keywords: Gemcitabine; Cisplatin; Bladder; radical nephroureterectomy; ureterectomy; 10-208
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — Gemcitabine; Cisplatin

ARMS (1):
- Gemcitabine and Cisplatin (Experimental): This is a Phase II Study of Gemcitabine and Cisplatin (GC) as neoadjuvant chemotherapy in patients with upper tract high-grade urothelial carcinoma who are candidates for radical nephroureterectomy or distal ureterectomy.
  Interventions: Drug: Gemcitabine and Cisplatin

INTERVENTIONS:
Drug: Gemcitabine and Cisplatin — Patients will receive four cycles of GC administered every 21 days. Gemcitabine 1,000 mg/m2 and Cisplatin 35 mg/m2 will be administered intravenously on days 1 and 8. A total of four cycles of therapy will be administered at 21 day intervals followed by radical nephroureterectomy or distal ureterectomy.

SUMMARY:
The purpose of this study is to see if getting chemotherapy with Gemcitabine and Cisplatin for four 21 day cycles for a total of 12 weeks can help shrink the tumor before undergoing surgery for kidney cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed high-grade upper tract transitional cell carcinoma at MSKCC or a participating site and/or radiographically visible tumor stage T2-T4a N0/X M0 disease with positive selective urinary cytology or high-grade concomitant bladder tumor. Hydronephrosis associated with tumor on biopsy will be considered invasive by definition.
* Medically appropriate candidate for radical nephroureterectomy or ureterectomy as per MSKCC or a participating site attending urologic oncologist
* Karnofsky Performance Status ≥ 70%
* Age ≥ 18 years of age
* Required Initial Laboratory Values:

  * Absolute neutrophil count ≥ 1500 cells/mm3
  * Platelets ≥ 100,000 cells/mm3
  * Hemoglobin ≥ 9.0g/dL
  * Bilirubin ≤ 1.2
  * Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 x ULN for the institution
  * Alkaline phosphatase ≤ 2.5 x ULN for the institution
  * Serum creatinine ≤ 1.3 mg/dL if male or ≤ 1.1 mg/dL if female OR calculated creatinine clearance ≥ 55 ml/min/1.73m^2 If female of childbearing potential, serum pregnancy test is negative.
* Patients with reproductive potential must use an effective method to avoid pregnancy for the duration of the trial.

ml/min/1.73m2 using the formula: CKD epi : GFR = 141 X min(Scr/κ,1)α X max(Scr/κ,1)-1.209 X 0.993Age X 1.018 [if female] X 1.159 [if black]

* Scr is serum creatinine, k is 0.7 for females and 0.9 for males, a is -0.329 for females and -0.411 for males, min indicates the minimum of Scr/k or 1, and max indicates the maximum of Scr/k or 1.
* If female of childbearing potential, serum pregnancy test is negative.
* Patients with reproductive potential must use an effective method to avoid pregnancy for the duration of the trial

Exclusion Criteria:

* Concomitant bladder urothelial carcinoma is acceptable if it is organ confined and surgically resectable.
* Presence of carcinoma in situ (CIS)
* Prior systemic chemotherapy (prior intravesical therapy is allowed)
* Prior radiation therapy to the bladder
* Evidence of NYHA functional class III or IV heart disease.
* Serious intercurrent medical or psychiatric illness, including serious active infection.
* Preexisting sensory grade 3 neuropathy
* Major surgery or radiation therapy < 4 weeks of starting study treatment.
* Concomitant use of any other investigational drugs
* Any of the following within the 6 months prior to study drug administration:

myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, or pulmonary embolism.

* Ongoing cardiac dysrhythmias of NCI CTCAE Version 4.0 grade ≥ 2.
* Uncontrolled hypertension (>150/100 mmHg despite optimal medical therapy).
* Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness or other active infection. Patients with HIV but no evidence of AIDS will be considered candidates.
* Concurrent treatment on another clinical trial involving an intervention which may affect the primary endpoint. Supportive care trials or non-treatment trials, e.g. QOL, are allowed.
* Ongoing treatment with therapeutic doses of warfarin or low molecular weight heparin (low dose warfarin up to 2 mg po daily or use of subcutaneous low molecular weight heparin for thromboembolic prophylaxis is allowed).
* Pregnancy or breast-feeding. Patients must be surgically sterile or be postmenopausal, or must agree to use effective contraception during the period of therapy. The definition of effective contraception will be based on the judgment of the MSKCC and participating site PI. Male patients must be surgically sterile or agree to use effective contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2010-12-14 (Actual); Primary Completion 2025-08-06 (Actual); Study Completion 2025-08-06 (Actual)

PRIMARY OUTCOMES:
To define the pathologic response rate (<pT2) | The time to disease progression is measured from the time of initiation of chemotherapyuntil the first date that systemic recurrence is objectively documented.
  of neoadjuvant Gemcitabine and Cisplatin regimen in patients with upper tract high-grade urothelial carcinoma. And is defined as the absence of high-grade carcinoma (<pT2 disease) and the absence of microscopic lymph node metastases (N0) on the final nephroureterectomy specimen.

SECONDARY OUTCOMES:
To determine the time to disease progression | Time to progression is measured from the time of initiation of chemotherapy until the 1st date that systemic recurrence is objectively documented. Systemic recurrence for this trial is defined as either metastatic or local pelvic recurrence.
  will be estimated using the methods of Kaplan and Meier in patients with upper tract high-grade urothelial carcinoma with neoadjuvant GC followed by radical nephroureterectomy.
To determine overall survival of patients | 3 years
  will be estimated using the methods of Kaplan and Meier in patients with upper tract high-grade urothelial carcinoma treated with neoadjuvant GC followed by radical nephroureterectomy.
To evaluate the safety and tolerability | every 2 weeks per cycle
  of neoadjuvant Gemcitabine and Cisplatin in this setting. Toxicity will be graded according to the National Cancer Institute Common Toxicity Criteria version 4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Coleman, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (9):
- United States (9):
  - Mayo Clinic - Arizona, Scottsdale, Arizona
  - Hartford Hospital (Data Collection Only), Hartford, Connecticut
  - Memorial Sloan Kettering at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Consent and Follow-Up only), Uniondale, New York
  - Lehigh Valley Health Network (Data Collection Only), Allentown, Pennsylvania

REFERENCES:
- [Derived] Coleman JA, Yip W, Wong NC, Sjoberg DD, Bochner BH, Dalbagni G, Donat SM, Herr HW, Cha EK, Donahue TF, Pietzak EJ, Hakimi AA, Kim K, Al-Ahmadie HA, Vargas HA, Alvim RG, Ghafoor S, Benfante NE, Meraney AM, Shichman SJ, Kamradt JM, Nair SG, Baccala AA Jr, Palyca P, Lash BW, Rizvi MA, Swanson SK, Muina AF, Apolo AB, Iyer G, Rosenberg JE, Teo MY, Bajorin DF. Multicenter Phase II Clinical Trial of Gemcitabine and Cisplatin as Neoadjuvant Chemotherapy for Patients With High-Grade Upper Tract Urothelial Carcinoma. J Clin Oncol. 2023 Mar 10;41(8):1618-1625. doi: 10.1200/JCO.22.00763. Epub 2023 Jan 5. PMID 36603175
- [Derived] Hird AE, Magee DE, Cheung DC, Sander B, Sridhar S, Nam RK, Kulkarni GS. Neoadjuvant Versus Adjuvant Chemotherapy for Upper Tract Urothelial Carcinoma: A Microsimulation Model. Clin Genitourin Cancer. 2021 Apr;19(2):e135-e147. doi: 10.1016/j.clgc.2020.10.001. Epub 2020 Oct 13. PMID 33168398
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm